CLINICAL TRIAL: NCT06094530
Title: Clinical Evaluation of 18F-FAPI-RGD PET/CT for Imaging of Fibroblast Activation Protein and Integrin avb3 in Various Tumor Types
Brief Title: 18F-FAPI-RGD PET/CT in Various Tumor Types
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-cancers
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical feasibility of 18F-FAPI-RGD PET/CT will be evaluated in 100 patients with various types of tumor, and the results will be compared with those of 18F-FDG.

DETAILED DESCRIPTION:
The aim of this study is to evaluate, in patients with various types of tumor, the radiotracer uptake and clinical feasibility of 18F-FAPI-RGD PET/CT compared with those of 18F-FDG PET/CT. To evaluate the diagnostic performance of 18F-FAPI-RGD and 18F-FDG PET imaging, the results of the visually interpreted PET images will be compared with the histopathologic results (via surgery or biopsy), which are used as the gold standard for the ﬁnal diagnosis. For patients for whom tissue diagnosis is not applicable, clinical and radiographic follow-up data will be used as the reference standard to validate the PET/CT ﬁndings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected or diagnosed tumors

Exclusion Criteria:

* Hypertension that is difficult to control with medication, and systolic blood pressure exceeding 160mmHg
* Complicated with chronic liver disease, myocardial infarction, stroke
* Female patients who are pregnant (or attempting to become pregnant within six months), breastfeeding, or unwilling to use contraception
* Abnormal cardiopulmonary function or mental state, unable to tolerate prone lying for 20 minutes

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically suspected or diagnosed tumors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of 18F-FAPI-RGD and 18F-FDG Uptake in Patients with different Tumors | 1 month
  Tracer uptake in normal organs (background) is quantiﬁed by SUVmean, which is delineated with a sphere that had a diameter of 1 cm (for small organs, including thyroid, salivary gland, and pancreas) to 2 cm(for other organs, including brain, heart, liver, kidney, spleen, muscle, and bone marrow) placed inside the organ parenchyma. The tumor-to background ratio (TBR) is calculated as tumor SUVmax/background SUVmean.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Doctor, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China